CLINICAL TRIAL: NCT06249620
Title: A Randomized Controlled Trial of Oral Suplementation With AM3, Hesperidin and Spermidine on Immunity Response and Biological Age in Healthy Volunteers.
Brief Title: Oral Supplementation With AM3, Hesperidin and Spermidine Supplementation on Immunity Response and Biological Age.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: P21110b
Record Dates: First submitted 2023-07-25; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: AM3; Biological age; Inmunology clock; Spermidine; Hesperidin
MeSH Terms: interventions — Immunoferon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): The product (with the active ingredients) is randomly given to 20 participants for ingestion for two months.The dosage regimen is two capsules per day in a single dose.
  Interventions: Dietary Supplement: Inmunoferon
- Placebo (Placebo Comparator): The other 20 participants will receive a similar looking product but with inert substances (placebo group).The dosage regimen is two capsules per day in a single dose.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inmunoferon — The dosage regimen is two capsules (with the active ingredients) per day in a single dose.The study lasted 8 weeks, with 2 interventional visits at baseline and at 8 weeks. Blood samples are collected twice: once on day 0 of the study and again at the final visit.
  Arms: Active group
Dietary Supplement: Placebo — The dosage regimen is two capsules (with inert ingredients) per day in a single dose.The study lasted 8 weeks, with 2 interventional visits at baseline and at 8 weeks. Blood samples are collected twice: once on day 0 of the study and again at the final visit.
  Arms: Placebo

SUMMARY:
The goal of this interventional study is to know the immune status of healthy participants and to obtain their biological age before and after two months of ingesting a dietary supplement. These individuals are compared with others who will be given a product of similar appearance, but without containing active components, being the constituents of the placebo group.

The study has a duration of 8 weeks, with 2 interventional visits (complete blood samples will be collected) at baseline and at 8 weeks.

In order to be included in the trial, the patient must read the Patient Information Sheet and sign the informed consent form.

The dosage regimen is two capsules per day in a single dose.

DETAILED DESCRIPTION:
Forty consenting volunteers will be included in this prospective, randomized, double-blind study and will be randomized by a statistician independent of the research team.

The study consists of two milestones, in which different parameters are evaluated to finally reach the main goal, to measure their immune status and their biological age after taking the supplement (whose active ingredients include AM3, polyamines and flavonoids):

- Complete blood samples are collected from participants at milestone 1. To determine immune functions; neutrophils, lymphocytes and NK cells are measured. The adherence and chemotaxis capacity of neutrophils and lymphocytes is determined, as well as neutrophil phagocytosis and lymphocyte proliferation. In addition, the release of pro-inflammatory and anti-inflammatory cytokines is assessed.

In parallel, each participant will be given a survey to assess their perception of stress, which they will have to complete before and after 2 months of ingestion of the product (experimental and placebo).

- In milestone 2, oxidative and inflammatory stress parameters are analyzed. Regarding oxidative stress: catalase activity, glutathione reductase activity and reduced glutathione concentration are measured. In terms of inflammatory stress: concentrations of both proinflammatory and anti-inflammatory cytokines released are measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who give their consent for the study will be included after having read and understood the information provided in the informed consent document
* Between 29-65 years old
* Residents in the Community of Madrid

Exclusion Criteria:

* Volunteers with no allergies or intolerances to the product
* Patologies
* Excessive alcohol consumption
* Pregnant women
* Antioxidants intake from supplements

Ages: 29 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Biological Age | Baseline and Week 8
  The Biological Age will be determined at baseline and week 8, by using the mathematical model 'Immunity Clock', based on the the natural killer activity, Lymphoproliferation and phagocytosis, and neutrophils and lymphocyts chemotaxis

SECONDARY OUTCOMES:
Change in catalase activity with the use of a spectrophotometer | Baseline and week 8
  Measuring catalase activity with the use of a spectrophotometer will be used to assess oxidative stress at baseline and week 8 of treatment.
Change in Glutathione peroxidase levels | Baseline and week 8
  To determine glutathione peroxidase levels at baseline and week 8 to asseess oxidative stress.
Change in Glutathione reductase levels | Baseline and week 8
  To determine glutathione reductase levels at baseline and week 8 to assess oxidative stress.
Change in reduced/oxized glutathione concentrations (GSH/GSSG) | Baseline and week 8
  To determine educed/oxized glutathione concentrations at baseline and week 8 to asseess oxidative stress.
Change in inflammatory and anti-inflammatory cytokines levels | Baseline and week 8
  To determine levels of both inflammatory and anti-inflammatory cytokines at baseline and week 8 for evaluation of inflammatory stress.
Change in Malondialdehyde concentrations | Baseline and week 8
  To determine concentration levels of malondialdehyde at baseline and at week 8 to evaluate peroxidative damage.
Change in neutrophil levels | Baseline and week 8
  To determine neutrophil levels at baseline and week 8 to analyze the immunological functions.
Change in lymphocyte levels | Baseline and week 8
  To determine lymphocite levels at baseline and week 8 to analyze the immunological functions.
Change in cytotoxic activity of natural killer | Baseline and week 8
  The cytotoxic activity of NK cells was assessed by colorimetry of target cell lysis at baseline and week 8 of tretment to analyze the immunological functions.
Change in chemotaxis index | Baseline and week 8
  To analyze the immunological functions, the chemotaxis index was calculated at baseline and week 8 to assess the migration capacity of neutrophils and lymphocytes .
Change in lymphoproliferation levels | Baseline and week 8
  To analyze the immunological functions, lymphoproliferation capacity by neutrophils was measured at baseline and week 8.
Change in phagocytosis activity | Baseline and week 8
  To analyze the immunological functions, phagocytosis activity by the neutrophils will also be determined at baseline and week 8 of treatment.
  Phagocytosis is a critical biological activity through which the host can protect itself from infectious and non-infectious environmental particles and remove unwanted host cells in order to maintain tissue homeostasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Biología Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wayne SJ, Rhyne RL, Garry PJ, Goodwin JS. Cell-mediated immunity as a predictor of morbidity and mortality in subjects over 60. J Gerontol. 1990 Mar;45(2):M45-8. doi: 10.1093/geronj/45.2.m45. PMID 2313042
- [Result] De la Fuente M, Miquel J. An update of the oxidation-inflammation theory of aging: the involvement of the immune system in oxi-inflamm-aging. Curr Pharm Des. 2009;15(26):3003-26. doi: 10.2174/138161209789058110. PMID 19754376
- [Result] Foreman KJ, Marquez N, Dolgert A, Fukutaki K, Fullman N, McGaughey M, Pletcher MA, Smith AE, Tang K, Yuan CW, Brown JC, Friedman J, He J, Heuton KR, Holmberg M, Patel DJ, Reidy P, Carter A, Cercy K, Chapin A, Douwes-Schultz D, Frank T, Goettsch F, Liu PY, Nandakumar V, Reitsma MB, Reuter V, Sadat N, Sorensen RJD, Srinivasan V, Updike RL, York H, Lopez AD, Lozano R, Lim SS, Mokdad AH, Vollset SE, Murray CJL. Forecasting life expectancy, years of life lost, and all-cause and cause-specific mortality for 250 causes of death: reference and alternative scenarios for 2016-40 for 195 countries and territories. Lancet. 2018 Nov 10;392(10159):2052-2090. doi: 10.1016/S0140-6736(18)31694-5. Epub 2018 Oct 16. PMID 30340847
- [Result] Medvedev ZA. An attempt at a rational classification of theories of ageing. Biol Rev Camb Philos Soc. 1990 Aug;65(3):375-98. doi: 10.1111/j.1469-185x.1990.tb01428.x. No abstract available. PMID 2205304
- [Result] HARMAN D. Aging: a theory based on free radical and radiation chemistry. J Gerontol. 1956 Jul;11(3):298-300. doi: 10.1093/geronj/11.3.298. No abstract available. PMID 13332224
- [Result] Martinez de Toda I, Mate I, Vida C, Cruces J, De la Fuente M. Immune function parameters as markers of biological age and predictors of longevity. Aging (Albany NY). 2016 Nov 28;8(11):3110-3119. doi: 10.18632/aging.101116. PMID 27899767
- [Result] Martinez de Toda I, Vida C, Diaz-Del Cerro E, De la Fuente M. The Immunity Clock. J Gerontol A Biol Sci Med Sci. 2021 Oct 13;76(11):1939-1945. doi: 10.1093/gerona/glab136. PMID 33979432
- [Result] Martinez de Toda I, Ceprian N, Diaz-Del Cerro E, De la Fuente M. The Role of Immune Cells in Oxi-Inflamm-Aging. Cells. 2021 Nov 1;10(11):2974. doi: 10.3390/cells10112974. PMID 34831197
- [Result] Arranz L, Fernandez C, Rodriguez A, Ribera JM, De la Fuente M. The glutathione precursor N-acetylcysteine improves immune function in postmenopausal women. Free Radic Biol Med. 2008 Nov 1;45(9):1252-62. doi: 10.1016/j.freeradbiomed.2008.07.014. Epub 2008 Jul 27. PMID 18694818
- [Result] Maggini S, Pierre A, Calder PC. Immune Function and Micronutrient Requirements Change over the Life Course. Nutrients. 2018 Oct 17;10(10):1531. doi: 10.3390/nu10101531. PMID 30336639
- [Result] Garrido A, Cruces J, Ceprian N, De la Fuente M. Improvements in Behavior and Immune Function and Increased Life Span of Old Mice Cohabiting With Adult Animals. J Gerontol A Biol Sci Med Sci. 2018 Jun 14;73(7):873-881. doi: 10.1093/gerona/gly043. PMID 29506242
- [Result] Rojo JM, Rejas MT, Ojeda G, Portoles P, Barasoain I. Enhancement of lymphocyte proliferation, interleukin-2 production and NK activity by inmunoferon (AM-3), a fungal immunomodulator: variations in normal and immunosuppressed mice. Int J Immunopharmacol. 1986;8(6):593-7. doi: 10.1016/0192-0561(86)90031-7. PMID 3491798
- [Result] Moya P, Baixeras E, Barasoain I, Rojo JM, Ronda E, Alonso ML, Portoles A. Immunoferon (AM3) enhances the activities of early-type interferon inducers and natural killer cells. Immunopharmacol Immunotoxicol. 1987;9(2-3):243-56. doi: 10.3109/08923978709035213. PMID 2449486
- [Result] Sanchez Palacios A, Garcia Marrero JA, Schamann F. [Immunologic clinical evaluation of a biological response modifier, AM3, in the treatment of childhood infectious respiratory pathology]. Allergol Immunopathol (Madr). 1992 Jan-Feb;20(1):35-9. Spanish. PMID 1509986
- [Result] Villarrubia VG, Valladolid JM, Elorza FL, Sada G, Vilchez JG, Jimenez M, Herrerias JM. Therapeutic response of chronic active hepatitis B (CAHB) to a new immunomodulator: AM3. Immunohematological effects. Immunopharmacol Immunotoxicol. 1992;14(1-2):141-64. doi: 10.3109/08923979209009217. PMID 1597653
- [Result] Villarrubia VG, Moreno Koch MC, Calvo C, Gonzalez S, Alvarez-Mon M. The immunosenescent phenotype in mice and humans can be defined by alterations in the natural immunity reversal by immunomodulation with oral AM3. Immunopharmacol Immunotoxicol. 1997 Feb;19(1):53-74. doi: 10.3109/08923979709038533. PMID 9049659
- [Result] Serrano-Gomez D, Martinez-Nunez RT, Sierra-Filardi E, Izquierdo N, Colmenares M, Pla J, Rivas L, Martinez-Picado J, Jimenez-Barbero J, Alonso-Lebrero JL, Gonzalez S, Corbi AL. AM3 modulates dendritic cell pathogen recognition capabilities by targeting DC-SIGN. Antimicrob Agents Chemother. 2007 Jul;51(7):2313-23. doi: 10.1128/AAC.01289-06. Epub 2007 Apr 23. PMID 17452477
- [Result] Martin-Vilchez S, Molina-Jimenez F, Alonso-Lebrero JL, Sanz-Cameno P, Rodriguez-Munoz Y, Benedicto I, Roda-Navarro P, Trapero M, Aragoneses-Fenoll L, Gonzalez S, Pivel JP, Corbi AL, Lopez-Cabrera M, Moreno-Otero R, Majano PL. AM3, a natural glycoconjugate, induces the functional maturation of human dendritic cells. Br J Pharmacol. 2008 Jun;154(3):698-708. doi: 10.1038/bjp.2008.87. Epub 2008 Apr 14. PMID 18414382
- [Result] Albillos A, Nieto M, Ubeda M, Munoz L, Fraile B, Reyes E, Lledo L, Blanco I, Pastor O, Salas C, Lario M, Monserrat J, Bataller R, Alvarez-Mon M. The biological response modifier AM3 attenuates the inflammatory cell response and hepatic fibrosis in rats with biliary cirrhosis. Gut. 2010 Jul;59(7):943-52. doi: 10.1136/gut.2008.168831. Epub 2010 May 4. PMID 20442198
- [Result] Yuan CL, Lin SW, Cheng MH. Inhibition of Molecular Signaling in Huh-7 Cells by AM3: A Novel Chemotherapeutic Agent for Hepatocellular Carcinoma. Med Chem. 2016;13(1):49-56. doi: 10.2174/1573406412666160622130036. PMID 27342078
- [Result] Fernandez-Lazaro D, Fernandez-Lazaro CI, Mielgo-Ayuso J, Adams DP, Garcia Hernandez JL, Gonzalez-Bernal J, Gonzalez-Gross M. Glycophosphopeptical AM3 Food Supplement: A Potential Adjuvant in the Treatment and Vaccination of SARS-CoV-2. Front Immunol. 2021 Jun 17;12:698672. doi: 10.3389/fimmu.2021.698672. eCollection 2021. PMID 34220861
- [Result] Larque E, Sabater-Molina M, Zamora S. Biological significance of dietary polyamines. Nutrition. 2007 Jan;23(1):87-95. doi: 10.1016/j.nut.2006.09.006. Epub 2006 Nov 20. PMID 17113752
- [Result] Ramani D, De Bandt JP, Cynober L. Aliphatic polyamines in physiology and diseases. Clin Nutr. 2014 Feb;33(1):14-22. doi: 10.1016/j.clnu.2013.09.019. Epub 2013 Oct 6. PMID 24144912
- [Result] Hesterberg RS, Cleveland JL, Epling-Burnette PK. Role of Polyamines in Immune Cell Functions. Med Sci (Basel). 2018 Mar 8;6(1):22. doi: 10.3390/medsci6010022. PMID 29517999
- [Result] Handa AK, Fatima T, Mattoo AK. Polyamines: Bio-Molecules with Diverse Functions in Plant and Human Health and Disease. Front Chem. 2018 Feb 5;6:10. doi: 10.3389/fchem.2018.00010. eCollection 2018. PMID 29468148
- [Result] Munoz-Esparza NC, Latorre-Moratalla ML, Comas-Baste O, Toro-Funes N, Veciana-Nogues MT, Vidal-Carou MC. Polyamines in Food. Front Nutr. 2019 Jul 11;6:108. doi: 10.3389/fnut.2019.00108. eCollection 2019. PMID 31355206
- [Result] Ramos-Molina B, Queipo-Ortuno MI, Lambertos A, Tinahones FJ, Penafiel R. Dietary and Gut Microbiota Polyamines in Obesity- and Age-Related Diseases. Front Nutr. 2019 Mar 14;6:24. doi: 10.3389/fnut.2019.00024. eCollection 2019. PMID 30923709
- [Result] Nakanishi S, Cleveland JL. Polyamine Homeostasis in Development and Disease. Med Sci (Basel). 2021 May 13;9(2):28. doi: 10.3390/medsci9020028. PMID 34068137
- [Result] Sagar NA, Tarafdar S, Agarwal S, Tarafdar A, Sharma S. Polyamines: Functions, Metabolism, and Role in Human Disease Management. Med Sci (Basel). 2021 Jun 9;9(2):44. doi: 10.3390/medsci9020044. PMID 34207607
- [Result] Negrel S, Brunel JM. Synthesis and Biological Activities of Naturally Functionalized Polyamines: An Overview. Curr Med Chem. 2021;28(17):3406-3448. doi: 10.2174/0929867327666201102114544. PMID 33138746
- [Result] Bravo-San Pedro JM, Senovilla L. Immunostimulatory activity of lifespan-extending agents. Aging (Albany NY). 2013 Nov;5(11):793-801. doi: 10.18632/aging.100619. PMID 24389041
- [Result] Madeo F, Eisenberg T, Pietrocola F, Kroemer G. Spermidine in health and disease. Science. 2018 Jan 26;359(6374):eaan2788. doi: 10.1126/science.aan2788. PMID 29371440
- [Result] Stacchiotti A, Corsetti G. Natural Compounds and Autophagy: Allies Against Neurodegeneration. Front Cell Dev Biol. 2020 Sep 22;8:555409. doi: 10.3389/fcell.2020.555409. eCollection 2020. PMID 33072744
- [Result] Soda K. Spermine and gene methylation: a mechanism of lifespan extension induced by polyamine-rich diet. Amino Acids. 2020 Feb;52(2):213-224. doi: 10.1007/s00726-019-02733-2. Epub 2019 Apr 19. PMID 31004229
- [Result] Zhang M, Wang H, Tracey KJ. Regulation of macrophage activation and inflammation by spermine: a new chapter in an old story. Crit Care Med. 2000 Apr;28(4 Suppl):N60-6. doi: 10.1097/00003246-200004001-00007. PMID 10807317
- [Result] Proietti E, Rossini S, Grohmann U, Mondanelli G. Polyamines and Kynurenines at the Intersection of Immune Modulation. Trends Immunol. 2020 Nov;41(11):1037-1050. doi: 10.1016/j.it.2020.09.007. Epub 2020 Oct 12. PMID 33055013
- [Result] Zhang H, Simon AK. Polyamines reverse immune senescence via the translational control of autophagy. Autophagy. 2020 Jan;16(1):181-182. doi: 10.1080/15548627.2019.1687967. Epub 2019 Nov 6. PMID 31679458
- [Result] Latour YL, Gobert AP, Wilson KT. The role of polyamines in the regulation of macrophage polarization and function. Amino Acids. 2020 Feb;52(2):151-160. doi: 10.1007/s00726-019-02719-0. Epub 2019 Apr 23. PMID 31016375
- [Result] Barreca D, Gattuso G, Bellocco E, Calderaro A, Trombetta D, Smeriglio A, Lagana G, Daglia M, Meneghini S, Nabavi SM. Flavanones: Citrus phytochemical with health-promoting properties. Biofactors. 2017 Jul 8;43(4):495-506. doi: 10.1002/biof.1363. Epub 2017 May 12. PMID 28497905
- [Result] Mas-Capdevila A, Teichenne J, Domenech-Coca C, Caimari A, Del Bas JM, Escote X, Crescenti A. Effect of Hesperidin on Cardiovascular Disease Risk Factors: The Role of Intestinal Microbiota on Hesperidin Bioavailability. Nutrients. 2020 May 20;12(5):1488. doi: 10.3390/nu12051488. PMID 32443766
- [Result] Xiong H, Wang J, Ran Q, Lou G, Peng C, Gan Q, Hu J, Sun J, Yao R, Huang Q. Hesperidin: A Therapeutic Agent For Obesity. Drug Des Devel Ther. 2019 Nov 12;13:3855-3866. doi: 10.2147/DDDT.S227499. eCollection 2019. PMID 32009777
- [Result] Tejada S, Pinya S, Martorell M, Capo X, Tur JA, Pons A, Sureda A. Potential Anti-inflammatory Effects of Hesperidin from the Genus Citrus. Curr Med Chem. 2018;25(37):4929-4945. doi: 10.2174/0929867324666170718104412. PMID 28721824
- [Result] Hajialyani M, Hosein Farzaei M, Echeverria J, Nabavi SM, Uriarte E, Sobarzo-Sanchez E. Hesperidin as a Neuroprotective Agent: A Review of Animal and Clinical Evidence. Molecules. 2019 Feb 12;24(3):648. doi: 10.3390/molecules24030648. PMID 30759833
- [Result] Li C, Schluesener H. Health-promoting effects of the citrus flavanone hesperidin. Crit Rev Food Sci Nutr. 2017 Feb 11;57(3):613-631. doi: 10.1080/10408398.2014.906382. PMID 25675136
- [Result] Estruel-Amades S, Massot-Cladera M, Perez-Cano FJ, Franch A, Castell M, Camps-Bossacoma M. Hesperidin Effects on Gut Microbiota and Gut-Associated Lymphoid Tissue in Healthy Rats. Nutrients. 2019 Feb 2;11(2):324. doi: 10.3390/nu11020324. PMID 30717392
- [Result] Camps-Bossacoma M, Franch A, Perez-Cano FJ, Castell M. Influence of Hesperidin on the Systemic and Intestinal Rat Immune Response. Nutrients. 2017 Jun 6;9(6):580. doi: 10.3390/nu9060580. PMID 28587283
- [Result] Homayouni F, Haidari F, Hedayati M, Zakerkish M, Ahmadi K. Hesperidin Supplementation Alleviates Oxidative DNA Damage and Lipid Peroxidation in Type 2 Diabetes: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Phytother Res. 2017 Oct;31(10):1539-1545. doi: 10.1002/ptr.5881. Epub 2017 Aug 14. PMID 28805022
- [Result] Li Y, Kandhare AD, Mukherjee AA, Bodhankar SL. Acute and sub-chronic oral toxicity studies of hesperidin isolated from orange peel extract in Sprague Dawley rats. Regul Toxicol Pharmacol. 2019 Jul;105:77-85. doi: 10.1016/j.yrtph.2019.04.001. Epub 2019 Apr 13. PMID 30991075
- See also: Oxidation and Inflammation in the Immune and Nervous Systems, a Link Between Aging and Anxiety — https://link.springer.com/referenceworkentry/10.1007/978-3-319-99375-1_115
- See also: Estrategias para enlentecer el envejecimiento en modelos de ratón y en humanos. Efectos sobre la longevidad y la edad biológica — https://eprints.ucm.es/id/eprint/72582/1/T43232.pdf